CLINICAL TRIAL: NCT00231621
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, One-year Study of the Efficacy and Safety of Topiramate in the Treatment of Obese Subjects With Dyslipidemia
Brief Title: A Study on Efficacy and Safety of Topiramate in Treatment of Obese Subjects With Dyslipidemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated prior to completion to focus on the development of a controlled release formulation.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003730
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Obesity; Hyperlipidemia; Hypertriglyceridemia
Keywords: Obesity; Dyslipidemia; Hyperlipidemia; Triglyceride; HDL; LDL; Diabetes
MeSH Terms: conditions — Obesity; Hyperlipidemias; Hypertriglyceridemia; Dyslipidemias; Diabetes Mellitus | interventions — Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to compare the efficacy and safety of daily topiramate versus placebo for the treatment of obese subjects with dyslipidemia.

DETAILED DESCRIPTION:
Topiramate is not approved for the treatment of obesity. Studies have shown that topiramate reduces weight in obese patients with or without Type 2 diabetes, and may have the adjunctive benefit of reducing triglyceride and cholesterol levels in these patients. This double-blind, placebo controlled study evaluates the long-term efficacy of topiramate for reduction of weight and triglyceride levels in obese patients with borderline to high hypertriglyceridemia, and the safety and tolerability of topiramate in this patient population. The study consists of four phases: 4-week enrollment (screening) phase, 8-week titration phase (topiramate dose will be increased from 16mg/day to the assigned dose), 52-week maintenance phase, and 6-week follow-up. Effectiveness of topiramate will be evaluated by multiple measurements such as change in body weight, body mass index, fasting serum triglyceride levels, cholesterol and other lipid profiles. Safety evaluations will include incidence/severity of adverse events, vital signs, clinical laboratory results. The hypothesis is that topiramate as compared to placebo will provide a greater percent reduction in body weight and in fasting serum triglycerides from Week 0 (baseline) to Week 60. After the initial 8-weeks titration phase, the patients will be randomized to receive either 96mg (48mg twice daily) or 192mg (96mg twice daily) topiramate or placebo (twice daily) by mouth for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A Body Mass Index (BMI) >= 27 kg/m^2 and <50 kg/m^2
* Stable weight at least four months prior to the first enrollment visit
* Diagnosis of dyslipidemia (serum triglycerides representative of mild to moderate hypertriglyceridemia and low HDL or high LDL)
* Patients on lipid lowering medication should be on monotherapy with the same drug for at least 4 months and on the same dose for at least 2 months prior to the first enrollment
* Female patients must be postmenopausal for at least 1 year, surgically incapable of childbearing, practicing abstinence, or practicing an acceptable method of contraception (requires negative pregnancy test)

Exclusion Criteria:

* Contraindication or hypersensitivity to topiramate
* Pregnancy, nursing or women who plan to become pregnant during the study
* Enrollment fasting triglycerides <175 or >= 1000 mg/dL, and/or LDL >= 190 mg/dL
* Hyperlipidemia secondary to known disease
* Other significant medical conditions such as cardiovascular or liver disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2001-05; Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Percent change in body weight and the percent change in fasting serum triglycerides from baseline (Week 0) to Week 60.

SECONDARY OUTCOMES:
Absolute change in body weight, body mass index, triglycerides, and absolute and percentage changes in cholesterol measures from baseline to Week 60. Safety evaluations throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Study on Efficacy and Safety of Topiramate in Treatment of Obese Subjects with Dyslipidemia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=542&filename=CR003730_CSR.pdf